CLINICAL TRIAL: NCT00001305
Title: Studies of Growth Deficiency and Growth Hormone Treatment in Children With Osteogenesis Imperfecta Types III and IV
Brief Title: Growth Hormone Therapy in Osteogenesis Imperfecta
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 920034; 92-CH-0034
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Results first posted 2019-01-29 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2017-05-19

CONDITIONS: Osteogenesis Imperfecta
Keywords: Osteogenesis Imperfecta
MeSH Terms: conditions — Osteogenesis Imperfecta | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Growth Hormone (Experimental): Treatment of children with types III and IV osteogenesis imperfecta with Humatrope
  Interventions: Drug: Humatrope

INTERVENTIONS:
Drug: Humatrope — Patients receive a subcutaneous injection.

SUMMARY:
Growth deficiency is a key feature of severe Osteogenesis Imperfecta (OI) and a frequent feature of mild to moderate forms of the disease. The reason that children with OI are short is not fully understood. We do know that details such as the number of fractures suffered or the type of OI do not fully explain the short stature of OI. Growth patterns have been defined for children with OI Types I, III, and IV. At about 12 months of age, children with Types III and IV OI demonstrate a predictable plateau of their linear growth rate. Type IV OI children begin to resume a normal growth rate at about age four to five years, but they will not "catch up" to a normal height, as they have "lost" a significant period of growth. The plateau usually continues for children with Type III OI. The reason for this growth plateau is unknown. There have been no studies which evaluate the growth of OI children in this age range. Our previous studies of growth in OI children have begun at age 5 years.

We have studied growth in OI children for the past 10 years. Different medications have been tried to both stimulate growth and improve bone density. Some children have responded to growth hormone (their growth rate increased by at least 50%) and some did not. The majority of children who did respond were Type IV. However, we need to carefully treat and study more children to try to determine which children will benefit from growth hormone medication.

The Goals of this Study Are:

1. We want to try to find a cause for the growth plateau common in types III and IV OI. Long-term, our goal is to develop a treatment to eliminate this plateau.
2. We want to see how long and how well OI bone will respond to growth stimulation.
3. We hope to find a "predictor" for who will respond to growth hormone and who will not, by measuring your child's endocrine and growth hormone function before receiving any growth hormone treatment.
4. We want to measure the effects of growth stimulation on bone density, and the quality of OI bone.
5. We want to see if there are long term benefits resulting from this treatment in the form of final adult height, trunk height, and possibly improved function of the respiratory system.

Median Subject Age (on p. 1 of webpage): 1-15 years (replaces 0-20)

DETAILED DESCRIPTION:
Growth deficiency is a cardinal feature of severe Osteogenesis Imperfecta (OI) and a frequent feature of mild to moderate forms of this disease. Despite the prevalence of short stature among people with OI, few studies have examined treatment options for this feature of OI. Recombinant human growth hormone (rGH) is a treatment for growth deficiency which we have investigated. In our initial studies we have found that many OI children are responsive to rGH especially those with type IV OI. The purpose of this protocol is to examine the effect of growth hormone treatment on linear growth of children with types III and IV OI and correlate growth responsiveness with growth hormone-somatomedin axis and histomorphometry parameters of OI bone.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients will be recruited with the goal of including at least 10 each of individuals with clinical/biochemical criteria of types III and IV OI who are between 3 and 8 years of age.

Height: Individuals with type III OI have severe short stature by definition; individuals with type IV OI recruited to the study will have height less than the 3rd percentile for age. All individuals will be required to furnish growth records, especially height and head circumference, from at least the preceding two years.

Long bone status: Participants must have radiographic evidence that long bone epiphyses have not yet fused. In addition, 60 degrees or greater angulation of a femur will exclude a child, pending surgical management or medical clearance.

Spine: Prospective participants will be evaluated for scoliosis and spinal compressions. Participants with scoliosis greater than 40 degrees will be excluded unless evidence is presented that the scoliosis has been stable for the prior two years. Participants with corrective rods in their spine will be excluded.

Neuro status: All patients will be co-enrolled in 97-CH-0064, and will be screened for Basilar Invagination through that protocol. Children who are initially screened by spiral CT scan with MRI confirmation and determined to have severe BI will be excluded from participation in this study. Severe BI is defined by NIH data as distortion of the angle between the pons and medulla and or compression of posterior fossa contents. We are only beginning to define the parameters of BI in this population, and we do not know why some children with BI progress in severity and some do not. Until those questions are answered, we feel it would not be prudent to stimulate growth in a child we know to have a severe form of BI at enrollment.

Pulmonary status: All children will be co-enrolled in 97-CH-0064, and will have pulmonary function testing through that protocol. Tests will be scheduled as required for that protocol; namely, PFTs every 2 years if normal, every year if abnormal.

EXCLUSION CRITERIA:

Patients who develop scoliosis greater than 40 degrees and/or patients who progress to severe basilar invagination during the study will be removed from the study. Failure to comply with the outlined procedures (blood draws, endocrine testing, bone biopsies, and visit schedule) is also a criterion for withdrawal from the protocol.

Patients who become pregnant.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 1991-11-05; Primary Completion 2017-05-19 (Actual); Study Completion 2017-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan C Marini, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Marini JC, Bordenick S, Heavner G, Rose S, Hintz R, Rosenfeld R, Chrousos GP. The growth hormone and somatomedin axis in short children with osteogenesis imperfecta. J Clin Endocrinol Metab. 1993 Jan;76(1):251-6. doi: 10.1210/jcem.76.1.8421094.
- [Background] Prockop DJ, Kivirikko KI. Heritable diseases of collagen. N Engl J Med. 1984 Aug 9;311(6):376-86. doi: 10.1056/NEJM198408093110606. No abstract available. PMID 6146097
- [Background] Rose SR, Municchi G, Barnes KM, Cutler GB Jr. Overnight growth hormone concentrations are usually normal in pubertal children with idiopathic short stature--a Clinical Research Center study. J Clin Endocrinol Metab. 1996 Mar;81(3):1063-8. doi: 10.1210/jcem.81.3.8772577.
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1992-CH-0034.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Growth Hormone: Treatment of children with types III and IV Osteogenesis Imperfecta with Growth Hormone Humatrope 0.06 mg/kg/day, 6 of 7 days per week
Period: Overall Study
Arm/Group | Growth Hormone
Started | 42
Completed | 42
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Growth Hormone
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 42
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 38
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Who Met Criteria of Increase in Growth Rate Since Baseline.
Description: The proportion of subjects who met the study criteria of at least 50% increase in growth rate since baseline.
Time Frame: 1 year
Population: The analyses included only those subjects who completed 1 year of study
Measure: Count of Participants; unit: Participants
Arm/Group | Growth Hormone
Number analyzed (Participants) | 42
Participants | 25

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Growth Hormone
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 1/42
Other Adverse Events (participants affected / at risk) | 4/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Growth Hormone (N=42)
Suicide attempt (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Growth Hormone (N=42)
Headache (Nervous system disorders) | 3 (3)
Reaction to preservatives (Immune system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-04-18): https://cdn.clinicaltrials.gov/large-docs/05/NCT00001305/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-18): https://cdn.clinicaltrials.gov/large-docs/05/NCT00001305/SAP_001.pdf